CLINICAL TRIAL: NCT02834676
Title: Retrospective Evaluation of Treatment of Chronic Pain Related to Cervical Disc Hernia Using Chemonucleolysis Substance
Brief Title: Clinical Effects of Gelified Ethanol Application in Cervical Disc Hernia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, Assistant Professor, Sakarya University
Other Study IDs: Sakarya Cervical
Record Dates: First submitted 2016-07-01; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: DiscoGel(R); gelified ethanol; percutaneous treatment; Oswestry Disability Index (ODI); Visual analog Scale (VAS); Neuropathic Pain Questionnaire (DN-4); cervical
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemonucleolysis by Gelified Ethanol: Patients visiting the pain clinic of the hospital who had cervical discogenic or radicular pain that did not resolve after the use of conventional therapy and ozone-oxygen therapy. Written informed consent was obtained from all participants.
  Interventions: Drug: Gelified Ethanol

INTERVENTIONS:
Drug: Gelified Ethanol — Pain relief with chemonucleolysis by using gelified ethanol regard to age, sex, ASA score, and complications.
  Other Names: DiscoGel

SUMMARY:
The aim of the study is to evaluate the clinical effects of Discogel® Radiopaque Gelified Ethanol as therapeutic substance for nucleolysis application in the patients with cervical disc hernia who had chronic pain and weakness on the neck, shoulders and arms.

DETAILED DESCRIPTION:
This is a retrospective, single-center study that is going to be conducted from November 2013 to May 2016 on patients visiting the pain clinic of the hospital who were treated with DiscoGel® for cervical discogenic or radicular pain that did not resolve after the use of conventional therapy and ozone-oxygen therapy.

Data collected from medical record forms and electronic medical record system of the hospital were used in the retrospective analysis of medical data with regard to age, gender, complications.

A resident who has not involved in the study interviewed each patient by telephone on the follow up to collect the related information.

ELIGIBILITY:
Inclusion Criteria:

* continuous radicular pain radiating to the upper limb, with a duration ≥8 weeks and an intensity >4/10 as rated by the patient on a visual analog scale (VAS)
* resistant to appropriate conservative treatment combining anti-inflammatory drugs and ozone-oxygen therapy, and confirmed by imaging with CT or MRI of a herniated disc putting pressure on a nerve root consistent with the clinical pain.

Exclusion Criteria:

* history of surgery at the cervical spine, contraindication to percutaneous chemonucleolysis (coagulopathy or infection), imaging results that did not support the clinical results, the presence of a herniated disc excluded or calcified on imaging, possible interference with pain evaluation due to any medical condition or treatment, involvement of incomplete data collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted from November 2013 to May 2016 on patients visiting the pain clinic who had cervical diskogenic or radicular pain that did not resolve after the use of conventional therapy and ozone-oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
DiscoGel technique for pain relief assessed by Statistical Package for the Social Sciences (SPSS) v22.0 | 1 month
  Statistical assessment of each patient was evaluated on time intervals before procedure, in the 1st month after procedure for Visual analogue scale (VAS) score for pain

SECONDARY OUTCOMES:
Assessment of degree of disability and estimating quality of life based on Oswestry Disability Index (ODI) score by SPSS v22.0 | 3 months
  Statistical assessment of each patient was evaluated on time intervals before procedure, in the 3rd months after procedure for ODI score
Assessment of degree of disability and estimating quality of life based on Oswestry Disability Index (ODI) score by SPSS v22.0 | 1 month
  Statistical assessment of each patient was evaluated on time intervals before procedure, in the 1st month after procedure for ODI score
DiscoGel technique for pain relief assessed by Statistical Package for the Social Sciences (SPSS) v22.0 | 3 months
  Statistical assessment of each patient was evaluated on time intervals before procedure, in the 3rd months after procedure for Visual analogue scale (VAS) score for pain

CONTACTS AND LOCATIONS:
Overall Officials: Serbülent G Beyaz, AssocProf, Principal Investigator — Clinical Chair
Locations (1):
- Sakarya University Research and Training Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellini M, Romano DG, Leonini S, Grazzini I, Tabano C, Ferrara M, Piu P, Monti L, Cerase A. Percutaneous injection of radiopaque gelified ethanol for the treatment of lumbar and cervical intervertebral disk herniations: experience and clinical outcome in 80 patients. AJNR Am J Neuroradiol. 2015 Mar;36(3):600-5. doi: 10.3174/ajnr.A4166. Epub 2014 Nov 13. PMID 25395657
- [Result] Theron J, Cuellar H, Sola T, Guimaraens L, Casasco A, Courtheoux P. Percutaneous treatment of cervical disk hernias using gelified ethanol. AJNR Am J Neuroradiol. 2010 Sep;31(8):1454-6. doi: 10.3174/ajnr.A1923. Epub 2010 Jan 6. PMID 20053805
- [Result] Stagni S, de Santis F, Cirillo L, Dall'olio M, Princiotta C, Simonetti L, Stafa A, Leonardi M. A minimally invasive treatment for lumbar disc herniation: DiscoGel(R) chemonucleolysis in patients unresponsive to chemonucleolysis with oxygen-ozone. Interv Neuroradiol. 2012 Mar;18(1):97-104. doi: 10.1177/159101991201800113. Epub 2012 Mar 16. PMID 22440607